CLINICAL TRIAL: NCT05213078
Title: Family Caregivers in Underserved Populations Providing Complex Cancer Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 20137; NCI-2020-11090 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 20137 (Other: City of Hope Medical Center); P30CA033572 (NIH)
Record Dates: First submitted 2020-12-10; First posted 2022-01-28 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Malignant Female Reproductive System Neoplasm; Stage 0 Lung Cancer AJCC v8; Stage I Lung Cancer AJCC v8; Stage IA1 Lung Cancer AJCC v8; Stage IA2 Lung Cancer AJCC v8; Stage IA3 Lung Cancer AJCC v8; Stage IB Lung Cancer AJCC v8; Stage II Lung Cancer AJCC v8; Stage IIA Lung Cancer AJCC v8; Stage IIB Lung Cancer AJCC v8; Stage III Lung Cancer AJCC v8; Stage IIIA Lung Cancer AJCC v8; Stage IIIB Lung Cancer AJCC v8; Stage IIIC Lung Cancer AJCC v8; Stage IV Lung Cancer AJCC v8; Stage IVA Lung Cancer AJCC v8; Stage IVB Lung Cancer AJCC v8
MeSH Terms: conditions — Lung Neoplasms | interventions — Early Intervention, Educational; Educational Status; Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Supportive Care (teaching intervention, questionnaire) (Experimental): Participants attend 2 teaching sessions with a research nurse. Participants also complete questionnaires at baseline, 3, and 7 weeks.
  Interventions: Other: Educational Intervention; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Other: Educational Intervention — Receive teaching intervention
  Other Names: Education for Intervention; Intervention by Education; Intervention through Education; Intervention, Educational
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This clinical trial develops and tests a model of family caregiver education focused on the role of underserved family caregivers as providers of complex care in the home. Cancer patients have symptoms from their cancer or treatment and are then supported by family caregivers at home with tasks requiring technical skill. Family caregivers are often asked to provide complex care whether it involves decisions about managing symptoms or providing technical care for ports/pumps, tubes, or devices. Family caregivers often are not given enough information on how to provide care for patients at home needing complex care. The results from this study may help researchers refine and improve the intervention for caregivers through future research for caregivers on a much larger scale.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Develop methods of assessing and supporting family caregiving skills in providing complex care.

II. Develop family caregiver (FCG) teaching materials and methods of instruction to enhance skills preparedness.

III. Pilot test the intervention in a cohort of underserved FCGs.

OUTLINE:

Participants attend 2 teaching sessions with a research nurse. Participants also complete questionnaires at baseline, 3, and 7 weeks.

ELIGIBILITY:
Inclusion Criteria:

* PATIENT: Diagnosis of any stage lung or gynecologic (gyn) cancer
* PATIENT: Read and understand English
* PATIENT: Requires either complex physical care or complex decision making regarding symptoms
* PATIENT: Age 18 years or older
* FCG: Designated by the patient as their caregiver
* FCG: Read and understand English
* FCG: Age 18 years or older
* FCG: Providing complex care and/or complex decision-making

Exclusion Criteria:

* Inability to read and understand English

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2020-07-15 (Actual); Primary Completion 2022-03-09 (Actual); Study Completion 2022-03-09 (Actual)

PRIMARY OUTCOMES:
Change in Family caregiver distress scale | up to 7 weeks
  Descriptive statistics will be used to summarize the distress scale. Analysis of variance (ANOVA) will be used to compare scores at the three points of baseline, 3 weeks, and 7 weeks.
Change in Quality of life (QOL) scale | Up to 7 weeks
  Descriptive statistics will be used to summarize the Caregiver QOL scale. ANOVA will be used to compare scores at the three points of baseline, 3 weeks, and 7 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Betty Ferrell, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States